CLINICAL TRIAL: NCT04661189
Title: The Cognitive and spOrt Virtual EPIC Training Study: Investigating the Effects of Home-based Exercise and Cognitive Training in Cardiovascular Diseases
Brief Title: The Cognitive and spOrt Virtual EPIC Training Study for Cardiovascular Diseases
Acronym: COVEPICARDIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Principal Investigator, Louis Bherer, Associate Scientific Director, Direction of Prevention, Montreal Heart Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ICM 2020-2785
Record Dates: First submitted 2020-12-03; First posted 2020-12-10 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Cardiovascular Diseases
Keywords: cardiovascular diseases; home-based exercise training; cognitive training; COVID-19; rehabilitation; cognition
MeSH Terms: conditions — Cardiovascular Diseases; COVID-19 | interventions — Exercise; Cognitive Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multidomain intervention (Experimental): The multidomain intervention will combine a remote monitoring of home-based cognitive training with physical exercise training for 6-month.
  Interventions: Behavioral: Physical exercise training; Behavioral: Cognitive training
- Physical exercise intervention (Experimental): The physical exercises intervention will include the remote monitoring of physical exercise training for 6-month.
  Interventions: Behavioral: Physical exercise training

INTERVENTIONS:
Behavioral: Physical exercise training — Participants will be encouraged to complete exercise training programs in the form of video capsules available via Facebook or Youtube, created by kinesiologists of the Montreal Heart Institut EPIC prevention center. The videos last about 15 minutes and include a warm-up of 3 to 5 minutes, followed a 10-minute training and finally a 2-minute cool-down period. The exercises on video do not require any equipment and integrate, depending on the video, aerobic, muscular strengthening, flexibility and/or balance exercises. Several intensities are described according to the participants' level. Participants will be invited to perform exercise sessions at least 5 times a week, and will be monitored weekly by phone by a member of the research team. The exercise sessions can be performed at home using the video training program, as well as in sports centre or outdoors. For each session, participants have to report its duration, intensity, and the nature of the activity via a follow-up agenda.
Behavioral: Cognitive training — Participants will be encouraged to perform sessions of cognitive training 3 times per week (30 minutes/session). Two of these sessions will involve computer or tablet-based attentional control training targeting dual-tasking, updating and working memory, as well as inhibition and switching. Difficulty of cognitive training will be tailored to participants' performances. The remaining session will consist of memory training. Participants will be instructed different mnemotechnic, as well as be taught about memory in aging in general. The memory training will be provided by videos capsules. To track adherence to cognitive training, participants will be asked to complete a journal and mark days and times where they took part in the various cognitive training sessions.
  Arms: Multidomain intervention

SUMMARY:
COVEPICARDIO trial is designed to document the effects of remote monitoring of physical exercise and home-based cognitive training on cognitive and physical functions in older adults with cardiovascular diseases.

DETAILED DESCRIPTION:
Cardiac rehabilitation is a class I level A recommendation with clinical benefits that are now well documented. Due to the COVID-19 pandemic, accessibility to rehabilitation services and exercise training programs are limited. Quarantine measures can induce collateral damages to cardiovascular and psychological health, in particular in clinical population. Cardiovascular diseases (CVD) are associated with cognitive deficits and increased risk of dementia later in life. Specifically for CVD, physical inactivity and excessive sedentary lifestyle induced by confinement decrease cardiorespiratory capacity, increase the risk of acute events and rehospitalization. Maintaining a minimum of physical activity during a health crisis is fundamental. In this context, our team has developed an innovative program of exercise and cognitive training at home. Considering the added benefits of combining cognitive training to physical exercise to further enhance health and cognition in seniors with CVD, this project also addresses the added benefits of a multidomain intervention combining a home-based physical exercise intervention with a cognitive training.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 50 and older
* Have access to internet
* Have access to a tablet (i.e., iPad or Android) or a computer
* Diagnostic of cardiovascular disease (stable chronic systolic or diastolic heart failure, atrial fibrillation, documented atherosclerotic disease).
* Able to do light to moderate aerobic exercice training
* With no contraindication to exercise training

Exclusion Criteria:

* Non-cardiopulmonary limitation to exercise (e.g., arthritis)
* Severe exercise intolerance
* Respiratory disease (e.g., asthma, COPD, COVID-19)
* Mini Mental Scale Examination (MMSE) telephone version lower than 19/23

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Change in general cognitive functioning | Baseline and post-intervention at 6 months
  Validated remote version of Montreal Cognitive Assessment
Change in executive functions | Baseline and post-intervention at 6 months.
  Validated remote version of Rey auditory verbal learning test, Trail Making Test, as well as Phonological and Semantic Fluency, Similarity, and Digit Span neuropsychological tests and iPad tests (Composite Z-score).
Change in processing speed | Baseline and post-intervention at 6 months
  Validated remote version of Rey auditory verbal learning test, Trail Making Test, as well as Phonological and Semantic Fluency, Similarity, and Digit Span neuropsychological tests and iPad tests (Composite Z-score).
Change in episodic memory | Baseline and post-intervention at 6 months
  Validated remote version of Rey auditory verbal learning test, Trail Making Test, as well as Phonological and Semantic Fluency, Similarity, and Digit Span neuropsychological tests and iPad tests (Composite Z-score).

SECONDARY OUTCOMES:
Change in Walking speed | Baseline and post-intervention at 6 months.
  4-meter walking test (m/s).
Change in Functional mobility | Baseline and post-intervention at 6 months
  Timed up and Go test (s).
Change in Balance performance | Baseline and post-intervention at 6 months
  Timed one-leg standing test (s)
Change in Lower limb muscles strength | Baseline and post-intervention at 6 months
  Timed Sit-to-Stand test (s).
Change in Cardiorespiratory fitness | Baseline and post-intervention at 6 months
  Matthews cardiorespiratory fitness questionnaire (the score is an estimation of individual VO2 max (ml.kg.min) and range from 15-50, with a higher score indicating a higher VO2max)

OTHER OUTCOMES:
Change in Quality-of-life | Baseline and post-intervention at 6 months.
  36-Item Short Form Health Survey (Scale ranges from 0-100, with a higher score indicating a better health status).
Change in Depressive symptomatology | Baseline and post-intervention at 6 months.
  Geriatric Depression Scale questionnaire (Score ranges from 0-30, with a higher score indicating larger depressive symptomatology).
Change in Anxiety | Baseline and post-intervention at 6 months.
  State-Trait Anxiety Inventory questionnaire (Score ranges from 20-80, with a higher score indicating higher anxiety)
Change in Perceived stress | Baseline and post-intervention at 6 months.
  Perceived Stress Scale questionnaire (Score ranges from 0-4, with 0 no stress,1 mild stress, 3 moderate stress and 4 severe)
Change in Repetitive negative thinking | Baseline and post-intervention at 6 months.
  Perseverative thinking questionnaire (Score ranges from 0-60, with a higher score indicating more repetitive negative thinking)
Change in Self-perceived resilience | Baseline and post-intervention at 6 months.
  Connor-Davidson Resilience Scale 10 questionnaire (Score ranges from 0-40, with a higher indicating better the resilience)
Change in Perceived social support | Baseline and post-intervention at 6 months.
  Lubben Social Network Scale questionnaire (Score ranges from 0-30, with a higher score indicating more social engagement).
Change in Social and community activities involvement | Baseline and post-intervention at 6 months.
  Social and community involvement questionnaire (Score ranges from 0-200, with a higher score indicating more social and community involvement).
Change in Self-reported physical activity | Baseline and post-intervention at 6 months.
  Physical Activity Scale for the Elderly questionnaire (Score ranges from 0-400, with a higher score indicating better level of physical activity).
Change in Sleep quality | Baseline and post-intervention at 6 months.
  Pittsburg Sleep Quality Index questionnaire (Score ranges from 0-21, with a higher score indicating worse sleep quality)
Change in Risk of sleep apnea | Baseline and post-intervention at 6 months.
  Berlin Questionnaire (Participants are classified into High Risk or Low Risk based on their responses to the individual items and their overall scores in the symptom categories.High Risk: if there are 2 or more categories where the score is positive. Low Risk: if there is only 1 or no categories where the score is positive).
Dietary patterns | Baseline
  Short Diet Questionnaire (Score ranges from 15-45 points, with a score between 15-29 categorised as unhealthy, 30-37 as somewhat unhealthy, and 38 or more as a healthy diet).
Intolerance of Uncertainty | Baseline
  Intolerance of Uncertainty scale questionnaire (Score ranges from 27-135, with a higher score indicating higher intolerance of uncertainty).
Anxiety Sensitivity | Baseline
  Anxiety Sensitivity Index questionnaire (Score ranges from 0-64, with a higher score indicating a higher sensitivity to anxiety)
Perceived vulnerability to disease | Baseline
  Perceived vulnerability to disease questionnaire (Score ranges from 15-95, with a higher score indicating a higher perceived vulnerability to disease).
Cognitive Reserve | Baseline
  Rami and colleagues' cognitive reserve questionnaire (Scale ranges from 0-26, with a higher score indicating a greater cognitive reserve).
Self-reported masculinity and femininity traits | Baseline
  Short Form Bem Sex-Role Inventory questionnaire (30 items questionnaire with 10 items assessing the femininity traits, 10 items assessing the masculinity traits, and 10 items neutral, not scored. Two scores are calculated for femininity and masculinity, respectively, and range from 10-70, whit a higher score indicating a higher femininity or masculinity trait).

CONTACTS AND LOCATIONS:
Locations (1):
- Preventive medicine and physical activity centre (centre EPIC), Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Besnier F, Dupuy EG, Gagnon C, Vincent T, Vrinceanu T, Blanchette CA, Iglesies-Grau J, Saillant K, Chabot-Blanchet M, Belleville S, Juneau M, Vitali P, Gayda M, Nigam A, Bherer L. Effects of home-based exercise with or without cognitive training on cognition and mobility in cardiac patients: A randomized clinical trial. Geroscience. 2025 Aug;47(4):5651-5667. doi: 10.1007/s11357-025-01530-y. Epub 2025 Feb 3. PMID 39899189
- [Derived] Besnier F, Dupuy EG, Gagnon C, Vincent T, Gregoire CA, Blanchette CA, Saillant K, Bouabdallaoui N, Grau JI, Berube B, Olmand M, Marin MF, Belleville S, Juneau M, Vitali P, Gayda M, Nigam A, Bherer L. Investigation of the Effects of Home-Based Exercise and Cognitive Training on Cognitive and Physical Functions in Cardiac Patients: The COVEPICARDIO Study Protocol of a Randomized Clinical Trial. Front Cardiovasc Med. 2021 Dec 6;8:740834. doi: 10.3389/fcvm.2021.740834. eCollection 2021. PMID 34938780